CLINICAL TRIAL: NCT05472714
Title: Integration of Multimodal Cancer Predisposition Genetic Counseling Practices Within the Pediatric Oncology Setting: Video Intervention for Newly Diagnosed Families Undergoing Genetic Testing
Brief Title: Educational Video for Genetic Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-019152; R21HG011912 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Genetic Disease; Cancer
Keywords: genetic testing; genetic counseling; germline testing; educational video
MeSH Terms: conditions — Genetic Diseases, Inborn; Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison between year 1 and year 2 cohorts, with year 2 cohort receiving intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without Video (No Intervention): In year 1, investigators will recruit families of patients receiving the current standard-of-care approach to tumor-normal genetic testing with provider based education.
- With Video (Experimental): In year 2, investigators will recruit families of patients receiving the updated standard-of-care approach to tumor-normal genetic testing with provider based education and an educational video.
  Interventions: Other: Educational Video

INTERVENTIONS:
Other: Educational Video — Investigators will develop an informational video to be presented within one week of diagnosis of a tumor to those referred for tumor normal paired genetic testing.
  Arms: With Video

SUMMARY:
Develop and evaluate the acceptability, feasibility, and preliminary efficacy of an informational video on paired tumor/normal testing for children and adolescents with a new diagnosis of cancer, tumors or other diagnosis.

DETAILED DESCRIPTION:
As over 15% of pediatric cancers are associated with a cancer predisposition, it is increasingly becoming standard of care for children with cancer, as well as those with suspected hereditary risk, to be evaluated for germline cancer predisposition. Unfortunately, the increase in pediatric genetic testing has exceeded the pace of research establishing best practices to optimize delivery of care for patients undergoing testing and their families. Tumor/normal genetic testing (testing of both tumor tissue and a paired normal sample) at time of cancer diagnosis or relapse is now widespread in pediatric oncology to improve cancer diagnostics, prognostics, and treatment; this testing also has potential to uncover underlying cancer predisposition syndromes with lifelong implications. Disseminating information at the time of cancer diagnosis is difficult, and is best done by a provider with expertise in cancer genetics. Thus, Investigators will develop an informational video for use prior to tumor/normal genetic testing to augment genetic counseling resources to support patients and families.

In this study, Investigators will develop and evaluate the acceptability, feasibility, and preliminary efficacy of an informational video on paired tumor/normal testing for children and adolescents with a new diagnosis of cancer, tumors or other diagnosis. Investigators will use a non randomized trial whereby a convenience sample of patients/families will be recruited to be controls in Year 1, followed by a convenience sample that will be allocated the video intervention In Year 2. To evaluate the impact of the video intervention, Investigators will compare assessments of two cohorts- an unexposed (no video intervention, Year 1) and exposed (video intervention, Year 2).

ELIGIBILITY:
Inclusion Criteria:

Parents

1. Parent or Legal Guardian of a patient with a new diagnosis of cancer, tumor, or other diagnosis referred for tumor/normal sequencing (proband) in the Cancer Center at the Children's Hospital of Philadelphia (CHOP)
2. Able to be approached within 1-4 weeks of tumor/normal sequencing
3. Appropriate to approach per oncology team
4. No cognitive impairment limiting ability to complete measures
5. Ability to read and speak English fluently

Adolescent/Young Adult (AYA) probands

1. Child proband receiving germline testing in the Cancer Center at CHOP
2. Ages 12+
3. Able to be approached within 1-4 weeks of tumor/normal sequencing
4. Appropriate to approach per oncology team
5. No cognitive impairment limiting ability to complete measures
6. Ability to read and speak English fluently

Exclusion Criteria:

1) Not meeting any of inclusion criteria.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
Knowledge Score - Before Results | up to 4 weeks after testing
  The primary outcome is the primary caregiver's knowledge score measured before receipt of genetic results. Knowledge score is a 12-point true/false questionnaire. Higher scores indicate higher genetic knowledge.

SECONDARY OUTCOMES:
Knowledge Score - After Results | Once, within 6 months after receipt of results
  The primary caregiver's knowledge score measured after receipt of genetic results, which is the same knowledge score measured before receipt of results. Knowledge score is a 12-point true/false questionnaire.
Knowledge Score - all caregivers and probands | Twice, prior to, and within 6 months after receipt of results
  Another secondary analysis will include data from all caregivers' (primary and secondary) and probands' (over 12 years of age) knowledge scores. The knowledge score is a 12-point true/false questionnaire.
Acceptability of use of an informational video on paired tumor/normal testing for participants with a new cancer or other diagnosis | One time, within 6 months after receipt of results
  Acceptability will be assessed using a questionnaire including a satisfaction with decision scale, a 6 question decision satisfaction measure, an impact of events scale for cancer-specific distress, a 15 item questionnaire, and a multidimensional impact of cancer risk assessment, a 6 item questionnaire.
Feasibility of an informational video on paired tumor/normal testing for children and adolescents with a new cancer diagnosis. | One time, within 6 months after receipt of results
  Feasibility will be assessed with absence of technical difficulties of video delivery and timeliness of delivery of video after recommendation for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne MacFarland, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators are committed to making all data, protocols, tools, and materials available to the scientific community, in compliance with Children's Hospital of Philadelphia policies and NIH "Sharing Data and Resources" statement, NIH Grants Policy Statement, and the NIH Office of Extramural Research, Division of Extramural Inventions & Technology Resources (DEITR) Intellectual Property Policy. This includes sharing of protocols freely with collaborators and sharing of data through peer-reviewed publication and presentation in scientific meetings. All members of the research team will comply with the NIH policy on sharing data by protecting the privacy and rights of human subjects involved in the research at all times. All members of the research team with comply with the Health Insurance Portability and Accountability Act of 1996 (HIPAA) and its accompanying regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Upon request